CLINICAL TRIAL: NCT06149507
Title: Effect of Acetaminophen Versus Ibuprofen in Treating Recurrent Apthous Ulcers in Pediatric Celiac Disease: A Randomized Pilot Study
Brief Title: Effect of Acetaminophen Versus Ibuprofen in Treating Recurrent Apthous Ulcers in Pediatric Celiac Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Afnan Osama Abdelnaby, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14422021417131
Record Dates: First submitted 2023-11-09; First posted 2023-11-29 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Celiac Disease in Children
MeSH Terms: interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen (Experimental): Syrup 10-15 mg/kg/dosage every 6-8 hours as needed and do not exceed more than 5 doses in 24 hours Duration 1 week
  Interventions: Drug: Acetaminophen
- ibuprofen (Active Comparator): Syrup 4-10 mg/kg/dosage every 4-6 hours as needed and do not exceed more than 5 doses in 24 hours Duration 1 week
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Acetaminophen — Prescribe the drug to the child
  Other Names: Paracetamol
  Arms: Acetaminophen
Drug: Ibuprofen — Prescribe the drug to the child
  Other Names: Brufin
  Arms: ibuprofen

SUMMARY:
Celiac disease (CD) is a chronic autoimmune enteropathy. It results from genetic predisposition and exposure to gluten-containing food. Individuals carrying human leucocytes antigen (HLA) markers DQ2 or DQ8 are genetically predisposed. Gluten is a protein found in wheat, rye, and barley; the main ingredients of bread, pasta, and pastries. Gluten works as a triggering factor for CD, but the interaction between genetic and environmental factors is still not fully understood.

Celiac disease can alter the absorption of drugs. Due to its vast surface area compared with the stomach, most drug absorption occurs in the small intestine and in celiac disease; the surface area available for absorption is substantially reduced due to villous atrophy.

Patients with celiac disease develop a variety of gastric disorders requiring oral medications, but the impact of damage to intestinal villi and other celiac disease squeal on drug absorption remains poorly understood. A review of the pertinent literature (English-language articles on research in adults published during the period 1970-August 2012) identified several reports of altered drug absorption mechanisms in patients with celiac disease, including accelerated or delayed gastric emptying, increased permeability of jejunal mucosa, changes in intraluminal pH, decreased intestinal surface area, and reduced intestinal cytochrome P-450 enzymes. A small number of published studies suggest that celiac disease may be associated with altered drug absorption, resulting in higher serum concentrations of propranolol, lower peak concentrations of acetaminophen and practolol, higher dosing requirements with levothyroxine, impaired or delayed absorption of certain antibiotics, and other pharmacokinetic effects with a potential impact on medication efficacy and toxicity. However, these studies involved very small patient samples and were poorly controlled, with some yielding contradictory results. More and larger pharmacokinetic studies in patients with celiac disease-especially studies of drugs that are dosed empirically or are not amenable to dosage adjustment according to vital signs or laboratory values-are needed.

DETAILED DESCRIPTION:
Celiac disease is an immune-mediated systemic disease triggered by intake of gluten in genetically susceptible individuals. The prevalence of celiac disease in the general population is estimated to be 1% in the world. Its prevalence differs depending on geographical and ethnic variations. The prevalence of celiac disease has increased significantly in the last 30 years due to the increased knowledge and awareness of physicians and the widespread use of highly sensitive and specific diagnostic tests for celiac disease.

Despite increased awareness and knowledge about celiac disease, up to 95% of celiac patients still remain undiagnosed. The presentations of celiac disease have significantly changed in the last few decades.

Classical symptoms of celiac disease occur in a minority of celiac patients, while older children have either minimal or atypical symptoms. Serologic tests for celiac disease should be done in patients with unexplained chronic or intermittent diarrhea, failure to thrive, weight loss, delayed puberty, short stature, amenorrhea, iron deficiency anemia, nausea, vomiting, chronic abdominal pain, abdominal distension, chronic constipation, recurrent aphthous stomatitis, and abnormal liver enzyme elevation, and in children who belong to specific groups at risk. Early diagnosis of celiac disease is very important to prevent long-term complications. Currently, the only effective treatment is a lifelong gluten-free diet. In this review, we will discuss the epidemiology, clinical findings, diagnostic tests, and treatment of celiac disease in the light of the latest literature.

When designing a clinical trial an appropriate justiﬁcation for the sample size should be provided in the protocol. This justiﬁcation could be based on formal power calculations or on other considerations such as the precision of the estimates of interest . However, there are a number of settings when designing a pilot investigation where there is no prior information upon which to base the sample size. For example, in phase I the study could be a bioavailability study for a new chemical entity, while for a later phase the study could be with a novel endpoint or in a previously unstudied group of patients (for the compound).

Of the four available studies of propranolol, two showed increased serum concentration levels in patients with celiac disease relative to those without celiac disease,12,23 one showed more rapid absorption with similar peak concentrations,24 and one showed no changes in peak concentrations or overall absorption but a reduction in jejunal absorption.22 Some inconsistencies in the results could be explained by slight differences in study protocols; specifically, the length of time study participants fasted before and after study drug administration, as well as variations in the temperature at which blood samples were stored (4C versus -20C) prior to testing, could have contributed to the dissimilarity of the results reported.

In general, it appears that some degree of altered absorption occurs with propranolol use in patients with celiac disease, but whether or not this translates to altered clinical outcomes is unknown and should be evaluated.

Until future trials studying these clinical effects directly, it may be prudent to initiate certain drugs at lower doses and implement dosage adjustments more cautiously in patients with celiac disease.

The earlier peak concentrations reported with aspirin and propranolol use and the increased overall AUC values reported for propranolol, cephalexin, clindamycin, sulfamethoxazole, trimethoprim, and methyldopa run counter to the general assumption that drug malabsorption occurs in patients

ELIGIBILITY:
Inclusion Criteria:

- 1. Children with clinical diagnosis with a celiac disease.

2. presence of recurrent apthous ulcers.

Exclusion Criteria:

* 1. History of allergy to any ingredient present in the drugs to be used for treatment.

  2. Children whose parents had no home or mobile phone to enable post-operative contact.

  3. Parent that who refuse to sign the informed consent.

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
change in pain intensity | 6 month
  faces pain scale score (from no pain [score 0] to maximum pain intensity [score 10] )

SECONDARY OUTCOMES:
presence of recurrent apthous ulcer | baseline, before intervention
  clinical observation complement by history from parents by yes or no
Occurrence of Dental enamel defects (DED) | baseline, before intervention
  Aine ' s classification of dental enamel defect score (0-4) dental enamel defects
Dental caries experience | baseline, before intervention
  CAST index (score"0: sound", "1: sealant", "2: restoration", "3: enamel lesions", "4,5: dentine lesions", "6: pulp involvement", "7: abscess/fistula", "8: tooth loss". if a situation did not match any code from 0 to 8, a code 9 was assigned.)
  l
Delayed dental eruption | baseline, before intervention
  number of teeth with delayed eruption

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elmotayam, PhD, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No